CLINICAL TRIAL: NCT00754754
Title: Brain Retraction Monitoring Sensor
Brief Title: Brain Retraction Monitoring Sensor Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Sponsor
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB 050960; BRI IFH 04.073
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Brain Surgery Requiring Significant Retraction of the Brain
Keywords: brain; surgery; retraction; injury; monitoring
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brain Retraction Monitoring Sensor (Experimental)
  Interventions: Procedure: Brain Retraction Monitoring Sensor

INTERVENTIONS:
Procedure: Brain Retraction Monitoring Sensor — This is a sensor incorporated into a brain retractor blade to monitor electrical activity and pressure applied to the brain during retraction required for the selected skull base operations.

SUMMARY:
The purpose of this study is to utilize a sensor incorporated into a brain retractor blade to monitor electrical activity and pressure applied to the brain during retraction required for the selected skull base operations. The overall goal of the study is to develop a protocol and guidelines to prevent the development of brain retraction injury during neurosurgical procedures requiring significant retraction.

DETAILED DESCRIPTION:
During neurosurgical operations for aneurysms, tumors, or other lesions located in the skull base, the surgeon must employ retracting devices in order to displace one or more lobes of the brain enough to gain adequate surgical exposure. These retractors are adjusted by hand to optimize exposure. It is often difficult for the surgeon to gauge the amount of pressure actually applied to the brain during such placement of the retractor. Moreover, it is also possible to position the blade of the retractor inadvertently such that a focal pressure point occurs at the tip of the retractor blade against the brain. Thus, injury to the brain can occur as a result of brain retraction when either the force applied is excessive or when the pressure is not adequately distributed to a large enough area of brain. This injury is thought to be the result of ischemia (inadequate blood flow) caused by the retraction, local trauma, or a combination of both. It has been estimated that this type of brain retraction injury occurs in approximately 10% of major cranial base tumor procedures or 5% of intracranial aneurysm surgeries. The specific aim of this research is to identify changes in electrical activity of brain tissue subjected to necessary retraction during neurosurgical procedures that may give forewarning of imminent brain retraction injury. It is anticipated that this information will permit development of guidelines that will enable the neurosurgeon to take steps to minimize such injury, i.e., by temporarily releasing or otherwise modifying the brain retraction. Cerebral electrical activity, together with the amount of retraction pressure being applied, will be recorded directly from the tissue at risk by means of a silastic electrode grid containing a pressure monitor placed on the surface of the cerebral cortex underneath the retractor blade.

ELIGIBILITY:
Inclusion Criteria:

* A patient must be scheduled to undergo skull base surgery requiring significant brain retraction
* Informed Consent

Exclusion Criteria:

* None, other than patients in whom major surgical complications are encountered that are unrelated to brain retraction may be excluded from subsequent data analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Duration and intensity of brain retraction pressure | Intraoperative

SECONDARY OUTCOMES:
Cortical DC potential | Postoperative
Local Electrocorticography (ECoG) | Postoperative
Radiographic retraction injury | Postoperative
Clinical deficits | Postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Ayad, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (3):
- United States (3):
  - Methodist Hospital, Indianapolis, Indiana
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Inova Fairfax Hospital, Falls Church, Virginia